CLINICAL TRIAL: NCT01081821
Title: A Double-blind, Placebo-controlled, Randomized, Single Ascending and Multiple Dose Study to Investigate the Safety and Pharmacokinetics of JNJ-39758979 in Healthy Japanese and Caucasian Adult Male Subjects
Brief Title: Single and Multiple Dose Study to Explore the Safety and Pharmacokinetics of JNJ-39758979 In Healthy Male Volunteers of Either Caucasian or Japanese Descent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016753
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: JNJ 39758979; Japanese descent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): single dose NJ-39758979/ matching placebo Single oral dose of JNJ-39758979 (either 50 100 300 600mg) or Placebo
  Interventions: Drug: single dose NJ-39758979/ matching placebo
- 002 (Experimental): multi-dose JNJ-39758979 /matching placebo JNJ-39758979 once daily oral dose for 14 days of 300 mg or Placebo
  Interventions: Drug: multi-dose JNJ-39758979 /matching placebo

INTERVENTIONS:
Drug: single dose NJ-39758979/ matching placebo — Single oral dose of JNJ-39758979 (either 50, 100, 300, 600mg) or Placebo
  Arms: 001
Drug: multi-dose JNJ-39758979 /matching placebo — JNJ-39758979 once daily oral dose for 14 days of 300 mg or Placebo
  Arms: 002

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and pharmacokinetics (how the drug is absorbed in the body, how it is distributed within the body and it is removed from the body over time) of single doses of JNJ-39758979 in healthy Japanese volunteers and multiple doses of JNJ-39758979 in healthy Japanese and Caucasian volunteers.

DETAILED DESCRIPTION:
This study will assess the safety and pharmacokinetics of JNJ-39758979 or placebo (which looks like the drug being studied but has no active ingredients) in healthy volunteers. This study is being conducted in two parts. Part 1 is a randomized (study drug will be assigned by chance), double-blind (neither the physician nor volunteer knows the identity of the assigned drug) study evaluating the safety, tolerability and pharmacokinetics of single doses of JNJ-39758979 and placebo in 36 healthy Japanese male volunteers. Part 2 is a randomized, double-blind study evaluating the safety, tolerability, and pharmacokinetics of multiple doses of JNJ-39758979 and placebo in 24 healthy Japanese males and 24 healthy Caucasian males. For Part 1, the participation period is a maximum of 56 days, including a screening visit, a 7-day in-clinic period and two follow-up visits. For Part 2, the participation period is a maximum of 202 days, including a screening visit, a 17-day in-clinic period and two follow-up visits. For both parts of the study, safety evaluations, which will include ECG (a cardiac function test), vital signs and monitoring of side-effects will be performed. Additionally, blood and urine samples will be collected for evaluation. Part 1: volunteers will receive a single oral (by mouth) dose of JNJ-39758979 (50, 100, 300, or 600mg) or placebo; Part 2: volunteers will receive an oral dose of JNJ-39758979 (300 mg) or placebo once a day for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Must be generally in good health
* If japanese, must have lived outside of Japan for no more than 5 years and whose parents and grandparents are Japanese
* Have negative result for HIV, hepatitis B, and hepatitis C
* Must be willing to use an acceptable method of birth control for 6 months after the last dose and to not donate sperm during the study and for 6 months after the last dose
* Must have a negative test for alcohol and drugs of abuse at check-in

Exclusion Criteria:

* History of alcohol or drug abuse within the last 5 years (consuming more than 14 drinks per week)
* Average consumption of more than 3 cups of caffeinated beverages (tea/coffee/cocoa/cola) per day
* Use of vitamins, herbal supplements, energy drinks or St.John's Wort (hypericin) for 14 days before first dosing
* Receipt of an experimental drug or medical device within the last month

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic and safety profile of single dose and multi-dose JNJ-39758979 as determined by lab and other safety evaluations | Through day 35 (after treatment) in Part 1 and through day 182 (after treatment) in Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Cypress, California, United States